CLINICAL TRIAL: NCT05409794
Title: Basal Plasma Lithium Levels and Suicidal Events (LIPS)
Brief Title: Basal Plasma Lithium Levels and Suicidal Events
Acronym: LIPS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL22_0039
Record Dates: First submitted 2022-06-03; First posted 2022-06-08 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Major Depressive Disorder; Suicidal Behavior; Bipolar Disorder
Keywords: Lithium; Depression; Suicide
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder; Depression; Suicide | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Suicide attempters/ideations: Patients currently suffering from a major depressive disorder and reporting at least one suicidal event (suicide attempt or hospitalization for suicidal ideation) over the last 12 months.
  Interventions: Biological: Blood sample
- Affective controls: Patients currently suffering from a major depressive disorder and reporting no suicidal event (suicide attempt or hospitalization for suicidal ideation) over the last 12 months.
  Interventions: Biological: Blood sample

INTERVENTIONS:
Biological: Blood sample — Blood sample for the determination of plasma lithium levels

SUMMARY:
Suicidal behavior is a major public health issue and there are currently no specific treatments for it.

However, lithium, the reference treatment for bipolar disorder, have been shown to be effective in preventing suicidal risk.

Apart from drug treatments, lithium is present in our environment and its levels varies from one individual to another, depending, especially, on diet.

Knowing that patients with a mood disorder generally have a poor lifestyle and a less rich and varied diet than the general population, variations in basal lithium levels can be expected in these patients.

DETAILED DESCRIPTION:
This study aims to assess the rate of depressed patients (unipolar or bipolar) with basal plasma lithium levels above 0.1 µeq/L.

It also aims to :

* compare basal plasma lithium levels according to the occurrence of a suicidal event in the year prior to inclusion ;
* assess the association of lithium levels with the intensity of current suicidal ideation ;
* assess the association of lithium levels with impulsiveness ;
* assess the association of lithium levels with characteristics of bipolar disorder (for patients with bipolar disorder) ;
* assess the association of lithium levels with emotional lability ;
* assess, in the patients with a suicidal event in the year prior to the inclusion, the association of lithium levels with the characteristics of suicide attempts

To do so, 158 patients currently suffering from a major depressive disorder and who have not received any lithium treatment over the last year, will be included and divided in two groups :

1. Depressed patients with a history of suicidal event over the last 12 months (suicide attempters/ideations) ;
2. Depressed patients with no history of suicidal event over the last 12 months (affective controls).

Following a clinical assessment, a blood sample will be collected from each participant to measure basal plasma lithium levels.

Study participation will be done in one day.

The investigators expect :

1. an inverse association between lithium levels and suicidal events in patients
2. an inverse association between lithium levels and impulsiveness and aggression in patients This study will contribute to a better knowledge on suicidal behavior, especially by confirming the protective effect of lithium and improving the understanding of the mechanisms involved.

This knowledge will eventually make it possible to develop prevention and management strategies.

More appropriate prevention and management strategies better adapted to patients at risk of suicide.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or over
* Current major depressive episode according to the DSM-5 (Diagnostic and Statistical Manual of Mental Disorders) criteria
* No lithium-based treatment over the last 12 months
* For suicide attempters/ideations only : suicidal event over the last 12 months
* For affective controls only : no suicidal event over the last 12 months

Exclusion Criteria:

* Lifetime diagnosis of schizoaffective disorder, schizophrenia or psychosis
* Pregnancy or breastfeeding
* Deprivation of freedom (by judicial or administrative decision)
* Legal protection measure (guardianship or curators)
* Inability to understand experimental procedures
* No affiliation to the French National Social Security System
* No consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients currently suffering from a major depressive disorder, with ot without a history of suicidal event over the last 12 months, seen in consultation or hospitalization in the Psychiatric Emergencies and Post Acute Care of Montpellier Univeristy Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 158 (Estimated)
Dates: Start 2022-12-09 (Actual); Primary Completion 2026-01-09 (Estimated); Study Completion 2027-01-09 (Estimated)

PRIMARY OUTCOMES:
Patients rate with lithium levels above 0.1 µeq/L | Baseline
  Rate of patients with basal plasma lithium levels, assessed at baseline, above the threshold of 0.1 µeq/L

SECONDARY OUTCOMES:
Basal plasma lithium levels | Baseline
  Basal plasma lithium levels (µeq/L) assessed in all participants at baseline.
Current suicidal ideation | Baseline
  Severity of current suicidal ideation, assessed with the Columbia Suicide Severity Rating Scale. The ideation severity subscale ranges from 1 to 5 (higher score indicating more severe ideation). The ideation intensity subscale includes 5 questions each ranging from 1 to 5 (higher score indication more intense ideation). The suicidal behavior subscale includes 4 yes/no questions. The suicidal behavior lethality subscale inquires about the level of actual or potential medical damage.
Impulsiveness level | Baseline
  Impulsiveness assessed with the Barratt Impulsiveness Scale (BIS). The total score ranges from 30 to 120 with a higher score indicating an increased impulsive behavior.
Aggression level | Baseline
  Aggression assessed with the 12 items Aggression Questionnaire (AQ-12). The questionnaire is divided in 4 subscales of 3 items (physical aggression, verbal aggression, anger, hostility) for each, the score ranges from 3 to 18 with a higher score indicating an increased aggressive behavior
Bipolar disorder characteristics | Baseline
  For patients with bipolar disorder (BD): type of BD, age of onset, rapid cycling over lifetime, number of manic/hypomanic/depressive episodes over lifetime and the last year.
Emotional lability | Baseline
  Emotional lability assessed with the Affective Lability Scale (ALS). The questionnaire is divided in 3 subscales (anxiety/depression, depression/elation and anger). For each subscale, higher score indicates an increased affective lability.
Suicide attempt characteristics | Baseline
  For patients with a suicide attempt in the year prior to inclusion : number of actual, aborted and interrupted suicide attempts, number of violent and serious attempts.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Montpellier, Montpellier, France